CLINICAL TRIAL: NCT05181631
Title: Diabetic/Metabolic Cardiomyopathy: Prevalence and Phenotype
Acronym: METAB-HEART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP210330
Record Dates: First submitted 2021-09-09; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-08

CONDITIONS: Cardiopathy; Diabetes; Metabolic Syndrome
Keywords: Cardiomyopathy; Diabetes; Obesity
MeSH Terms: conditions — Heart Diseases; Diabetes Mellitus; Metabolic Syndrome; Cardiomyopathies; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biobanking (Experimental): If the patient consents, two tubes of blood will be collected for biobanking, at the same time as routine tubes will be collected.
  Samples will be collected by hospital staff and stored following regulatory conditions of conservation in the biological resources center of Avicenne hospital .
  Interventions: Other: Biobanking

INTERVENTIONS:
Other: Biobanking — "Collection of blood (One tube of blood 4-5 ml + One EDTA tube of blood 5 ml) will be attempted for each participant at baseline. Availability of these samples will be indicated in the e-CRF.
  Samples will be collected by hospital staff and stored following regulatory conditions of conservation in CRB of Hospital Avicenne under the responsibility of Pr Marianne ZIOL. "

SUMMARY:
"Little is known about the prevalence, determinants and phenotypes of the cardiomyopathy associated with diabetes and/or metabolic syndrome. The emergence of new therapies (SGLT2 inhibitors) that may mitigate and even prevent the onset of heart failure offers new opportunities.The objective of this protocol is to evaluate the prevalence and phenotypes of cardiomyopathy confirmed by echography in people at high metabolic risk defined as living with diabetes or obesity."

DETAILED DESCRIPTION:
Heart failure (HF) is a frequent disease with a global prevalence of 2.3% that may culminate up to 10% in the elderly. HF is associated with poor outcomes, namely multiple recurrent hospitalizations and high mortality. It is well known for several decades that diabetes is associated with a high cardiovascular mortality, with most physicians initially focusing on coronary artery disease solely. More recently, the concept of specific diabetic and/or metabolic cardiomyopathy emerged with different phenotypes. Obesity and hypertension are highly prevalent in patients with type 2 diabetes (T2D) and several studies have shown similar "diabetic cardiomyopathies" and "obese cardiomyopathies". Congestive HF was found to be two to three times more frequent in patients with T2D than in those without. Asymptomatic HF is underestimated by lack of systematic screening of these patients which prevent them from benefiting from early therapeutics. To our knowledge, no previous study has been made with systematic screening for HF in obese patients without obvious HF signs. Several tools can be used to examine the possible presence of cardiomyopathy and/or HF. The detection of cardiomyopathy at an early, preclinical stage may be of particular interest. First, studies have demonstrated that HF management is more effective at an early stage, with some drugs being associated with a reverse remodeling. Second, the class of SGLT2 inhibitors has proven to reduce the risk of hospitalization for HF in high-risk patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years-old or more)
* At high metabolic risk: diabetes of any type and/or obesity (body mass index ≥ 30 kg/m²)
* Admission in the departement of Diabetology-Obesity-Nutrition, Avicenne Hospital, Bobigny, France
* Patient informed and having signed consent
* Patient affiliated to a social security scheme or entitled

Exclusion Criteria:

* Any know cardiac disease: coronary artery disease, heart failure, cardiomyopathy, pulmonary embolism < 6 months, pulmonary hypertension, rhythm disorders < 6 months
* Blood pressure > 180/110 mmHg
* Severe renal failure as defined by estimated glomerular filtration rate < 30 ml/min
* Age ≥ 80 years
* Previous inclusion in the study
* Patient under guardianship curatorship
* Patient on AME (aide médicale d'état)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2023-09-14 (Estimated)

PRIMARY OUTCOMES:
Echographic cardiomyopathy | 18 months
  Echographic cardiomyopathy defined as:
  * Reduced left ventricular ejection fraction (LVEF)<50%, and/or
  * Abnormal diastolic function defined as more than half of positive criteria among: E/e'>14, septal e' velocity<7cm/s or lateral e' velocity<10cm/s, Tricuspid regurgitation (TR) velocity>2.8m/s, indexed left atrial (LA) volume>34ml/m², and/or
  * Isolated left ventricular hypertrophy defined as LV mass ≥115g/m² in male and ≥95g/m² in female
  * Reduced contractility as defined by global longitudinal strain (GLS) < 20%, and/or If clinical sign & symptom, resting ECG and biomarkers are normal, then echography will not be carried out and the cardiomyopathy will be considered absent. "

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COSSON, Principal Investigator — Assistance Publique - Hôpitaux de Paris